CLINICAL TRIAL: NCT01810341
Title: SynapDx Autism Spectrum Disorder Gene Expression Analysis Study
Brief Title: SynapDx Autism Gene Expression Analysis Study (STORY)
Acronym: STORY
Status: Completed | Type: Observational
Sponsor: SynapDx (Industry)
Responsible Party: Sponsor
Other Study IDs: 12002
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Autism
Keywords: Autism; Autism Spectrum Disorders; RNA; Gene expression; Developmental Delay; Metabolites; DNA
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Development Group: In the Development Phase, analyses will be performed until the classification algorithm is finalized.
- Validation Group: The Validation Phase will assess the performance of the finalized classification algorithm in 300 subjects.

SUMMARY:
This study will prospectively enroll approximately 880 children, at least 18 months and less than 60 months of age, who have been referred to a pediatric developmental evaluation center. Enrolled children will have blood drawn for RNA gene expression analysis and optionally for metabolite, lipid and DNA analysis and undergo a clinical evaluation to determine the presence or absence of a diagnosis of ASD.

The primary objective of this study is:

- To develop an algorithm to classify blood RNA gene expression patterns to maximize agreement between the classification and a clinical assessment of presence or absence of Autism Spectrum Disorders (ASD).

The secondary objectives of this study are:

* To develop an algorithm to classify plasma metabolite and/or lipid profiles in such a way as to maximize agreement between the classification and a clinical assessment of presence or absence of ASD.
* To prospectively assess the clinical sensitivity and specificity of the plasma metabolite and/or lipid profile classification algorithm in a separate population consisting of children referred to a developmental evaluation clinic for a possible developmental disorder (DD).
* To evaluate clinical sensitivity and specificity of various combinations of gene expression signature, metabolite and/or lipid signatures, and presence of ASD-associated genetic variation detected by chromosomal microarray analysis (CMA) or sequencing protein-coding regions of the genome.

DETAILED DESCRIPTION:
The primary aim of this study is to define a gene expression signature indicative of ASD and to establish its clinical sensitivity and specificity. Clinician diagnosis of ASD will be made using DSM-5 as the reference standard instrument. The widely used diagnostic instrument Autism Diagnostic Observation Schedule (ADOS-2) is a typical component of the clinical assessment for a child diagnosed with ASD and this evaluation will be performed on all study participants. Secondary aims of this study are (1) to define metabolite and lipid signatures indicative of ASD and establish their clinical sensitivity and specificity and (2) to determine clinical sensitivity and specificity of various combinations of gene expression signature, metabolite and/or lipid signatures, and presence of ASD-associated genetic variation detected by CMA and sequencing protein-coding regions of the genome

Analyses: Details of the analysis will be specified in a Statistical Analysis Plan (SAP), which will include procedures for handling outliers, missing data, and differences across sites. The SAP will be reviewed and approved by a committee of Principal Investigators (PIs) before unblinding of the validation set.

Primary analyses: The primary outcomes of the study will be the estimates of the clinical sensitivity and specificity of the SDX-002 test to classify subjects according to DSM-5 ASD diagnosis, with associated 95% confidence intervals. Sensitivity and specificity will be assessed on the Validation Phase population based on agreement with the clinical diagnosis of presence or absence of Autism Spectrum Disorder by DSM-5 (published May 2013).

The gene expression signature will be trained on the 500 subject Development Phase set, using 5-fold cross validation over the results of several machine learning algorithms, including partial least squares, support vector machines, and boosted decision trees. The training procedure will generate estimated ROC curves for each method, as well as confidence intervals for the area under the curve (AUC). The final choice of a machine-learning algorithm will be based on AUC, as well as on the estimated performance at the chosen operating point on the ROC curve. The operating point will be chosen to provide high sensitivity at an acceptable specificity.

Secondary analyses: In the majority of patients enrolled to date, consent was obtained for collection of an optional bio-repository sample. The intended analysis of the bio-repository samples has now been established (see also, secondary objectives listed above). The metabolomic and lipomic signatures will be similarly assessed on the subset of the 500 subjects in the Development Phase set who consent to a bio-repository sample. In addition to the gene expression signature, metabolite and/or lipid signatures and DNA analysis will be combined with the gene expression signature in various configurations and the impact of these additional measures on clinical sensitivity and specificity will be evaluated. If these additional metabolomic/lipomic signatures and/or DNA analyses improve test performance, these elements may be included in the SDX-002 assay.

Sensitivity and specificity the final SDX-002 assay will also be assessed among subpopulations using demographic information and the results of developmental testing. There are likely to be few subjects in many of these subpopulations and caution will be used in interpreting the results. Planned subpopulation analyses include gender, age, ethnicity, ASD DSM-IV-TR diagnostic subcategory, DSM-5 ASD severity level (social communication and restricted interests/repetitive behaviors) and ADOS-2 scores.

ELIGIBILITY:
Inclusion Criteria:

* Referred to a developmental evaluation center for evaluation of a possible developmental disorder, other than isolated motor problems.
* At least 18 months and less than 60 months.
* Parent/legal guardian has been informed about the study and has signed an informed consent form.

Exclusion Criteria:

* Prior reliable diagnosis of Autism Spectrum Disorder (i.e. prior evaluation by a multi-disciplinary team has already reliably established Autism Spectrum Disorder diagnosis).
* Unable or unwilling to complete study procedures.

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 18 months to less than 60 months referred to a developmental evaluation center for evaluation of a possible developmental disorder.
Sampling Method: Probability Sample
Enrollment: 880 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
RNA gene expression in peripheral blood | Within 30 days of collection

SECONDARY OUTCOMES:
Metabolites, lipids and DNA variation in peripheral blood | Within 30 days of collection

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rathmell, MD, Study Director — SynapDx Corp
Locations (20):
- United States (18):
  - Melmed Center, Scottsdale, Arizona
  - Miller Children's Hospital, Long Beach, California
  - UC Davis MIND Institute, Sacramento, California
  - Emory University, Decatur, Georgia
  - Rush Medical Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Lurie Center Massachusetts General Hospital, Lexington, Massachusetts
  - Mount Sinai School of Medicine/Seaver Center, New York, New York
  - Institute for Behavioral Research on Staten Island, Staten Island, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Seattle Children's, Seattle, Washington
- Canada (2):
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario